CLINICAL TRIAL: NCT00674830
Title: Self-help Treatment for Insomnia in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Breast Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017738
Record Dates: First submitted 2008-05-07; First posted 2008-05-08 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): professionally administered cognitive-behavioral therapy
  Interventions: Behavioral: professionally administered cognitive-behavioral therapy
- 2 (Experimental): self-administered form of cognitive behavioral therapy
  Interventions: Behavioral: self-administered form of cognitive-behavioral therapy
- 3 (Placebo Comparator): usual care
  Interventions: Behavioral: placebo

INTERVENTIONS:
Behavioral: professionally administered cognitive-behavioral therapy — professionally administered CBT-I consisting of six weekly sessions
  Arms: 1
Behavioral: self-administered form of cognitive-behavioral therapy — self-administered CBT-I consisting of six short booklets and videotapes
  Arms: 2
Behavioral: placebo — usual care
  Arms: 3

SUMMARY:
The main goal of this population-based study is to assess the efficacy of two forms of cognitive-behavioral therapy (CBT) to treat various levels of insomnia symptoms in women with breast cancer: a professionally administered form and a patient self-administered form. It is hypothesized that the two treatment conditions will be associated with significantly greater improvements in sleep, psychological distress, fatigue, cognitive functioning, and quality of life, relative to the control condition (i.e., usual care). It is also hypothesized that the magnitude of effect sizes obtained in association with treatment at each time assessment will be greater for the professionally administered treatment than the self-administered treatment.

ELIGIBILITY:
Inclusion Criteria:

* To be receiving treatment for a diagnosis of breast or gynaecological cancer
* To obtain a score of 8 or higher on the Insomnia Severity Index (ISI) or to be using a hypnotic medication ≥ 1 night per week

Exclusion Criteria:

* To have received a diagnosis or being treated for :

  * a sleep disorder other than insomnia (e.g., sleep apnea)
  * a severe psychiatric disorder (e.g., psychotic disorder)
  * a severe cognitive disorder (e.g., dementia)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
sleep diary indices, actigraphy, Insomnia Severity Index | pre-treatment, post-treatment, 3 follow-up

SECONDARY OUTCOMES:
EORTC QLQ, MFI, CFQ, TCEIQ, HADS, DBAS, UHCSQ, costs | pre-treatement, post-treatment, 3 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Josée Savard, Ph.D., Principal Investigator — Centre de recherche de l'HDQ
Locations (1):
- Centre de recherche de l'HDQ, Québec, Quebec, Canada

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Savard J, Ivers H, Savard MH, Morin CM. Long-Term Effects of Two Formats of Cognitive Behavioral Therapy for Insomnia Comorbid with Breast Cancer. Sleep. 2016 Apr 1;39(4):813-23. doi: 10.5665/sleep.5634. PMID 26715229
- [Derived] Savard J, Ivers H, Savard MH, Morin CM. Is a video-based cognitive behavioral therapy for insomnia as efficacious as a professionally administered treatment in breast cancer? Results of a randomized controlled trial. Sleep. 2014 Aug 1;37(8):1305-14. doi: 10.5665/sleep.3918. PMID 25083010